CLINICAL TRIAL: NCT01073748
Title: The Effect of Paracetamol on Lower Airway Obstruction in Asthmatic Versus Non Asthmatic Children
Brief Title: The Effect of Single Dose Paracetamol on the Lower Airways of Asthmatic and Healthy Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Dr. Ruth Soferman, Tel-Aviv Sourasky Medical Center, Israel, Tel-Aviv Sourasky Medical Center, Israel
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: TASMC-10-RS-422-CTIL
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
Keywords: Asthma; Acetaminophen; paracetamol; FeNO; Spirometry; Lung function
MeSH Terms: conditions — Asthma | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- asthmatic subjects (Active Comparator): Asthmatic children will be randomly exposed to paracetamol and placebo consecutively and their lung functions will be blindly compared.
  Interventions: Drug: paracetamol
- Healthy children (Other): Children with no asthma as control group.
  Interventions: Drug: paracetamol

INTERVENTIONS:
Drug: paracetamol — single dose of paracetamol 15mg/kg.
  Other Names: Acetaminophen; Acamol

SUMMARY:
Asthma is a common inflammatory airway disease. Several researches have demonstrated a possible connection between asthma and exposure to paracetamol.

Our hypothesis is that even a single dose of paracetamol is sufficient to cause a measurable change in lung functions.

This trial aims to identify a possible effect of single dose paracetamol on lower airway function.

DETAILED DESCRIPTION:
Asthma is a common inflammatory airway disease and its prevalence is on the rise all around the world, Most significantly in children under 5 years.

Paracetamol is one of the most common drugs used with children at thus age groups and several studies have proved a causative connection between exposure to paracetamol and asthma prevalence as well as other allergic conditions.

The mechanism is presumably by reduction of glutathione level, resulting in oxidative burst and formation of reactive oxygen species (ROS).

In addition, paracetamol maybe directly cytotoxic to pneumocytes if given in overdose.

The goal of this research is to identify and quantify the effect of single dose of paracetamol on lung functions of asthmatic and healthy subjects.

The study group will include 40 children aged 7-16 years, who are known to have asthma and a control group of 20 healthy children.

The children will be randomized to receive a dose of paracetamol or placebo, and lung functions will be measured by both spirometry and Fraction of expired Nitric Oxide (FeNO) test.

Each child will receive both paracetamol and placebo, randomly in to consecutive tests, thus children will serve as their own control.

ELIGIBILITY:
Inclusion Criteria:

* age: 7-16 years
* research group: children who have been diagnosed as asthmatic according to the American thoracic society (ATS) criteria
* control group: children who are not known to have asthma

Exclusion Criteria:

* paracetamol sensitivity
* children with any kind of chronic disease (except asthma)
* children with non asthma related chronic lung disease
* acute asthma attack
* children on systemic steroids

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
A measurable change in lung functions in response to paracetamol exposure. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Soferman, M.D, Principal Investigator — TASMC
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel